CLINICAL TRIAL: NCT05636150
Title: A Phase II Clinical Study to Evaluate the Efficacy and Safety of Fuquinitinib Combined With S-1 in the Treatment of Patients With Advanced Esophageal Squamous Cell Carcinoma
Brief Title: A Phase II Clinical Study of Fruquintinib Combined With S-1 for Advanced Esophageal Squamous Cell Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Lin Zhao, chief physician, Peking Union Medical College Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-013-CH07 IIT-EC
Record Dates: First submitted 2022-11-23; First posted 2022-12-05 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2022-12

CONDITIONS: Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — HMPL-013; S 1 (combination)

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fruquintinib plus S-1 (Experimental): Cohort A: Fruquintinib 3 mg QD, oral dosing, 2 weeks on/1 weeks off+ S-1 40-60mg/time bid po d1-14 q3w.
  Cohort B: Fruquintinib 4 mg QD, oral dosing, 2 weeks on/1 weeks off+ S-1 40-60mg/time bid po d1-14 q3w.
  Cohort C: Fruquintinib 5 mg QD, oral dosing, 2 weeks on/1 weeks off+ S-1 40-60mg/time bid po d1-14 q3w.
  Interventions: Drug: Fruquintinib in Combination with S-1

INTERVENTIONS:
Drug: Fruquintinib in Combination with S-1 — Cohort A: Fruquintinib 3 mg QD, oral dosing, 2 weeks on/1 weeks off+ S-1 40-60mg/time bid po d1-14 q3w.
  Cohort B: Fruquintinib 4 mg QD, oral dosing, 2 weeks on/1 weeks off+ S-1 40-60mg/time bid po d1-14 q3w.
  Cohort C: Fruquintinib 5 mg QD, oral dosing, 2 weeks on/1 weeks off+ S-1 40-60mg/time bid po d1-14 q3w.
  Patients will be treated until disease progression, death, unacceptable toxicity, loss of follow-up, withdrawal of consent or other conditions meet the end of treatment criteria.

SUMMARY:
Investigators conduct the clinical trial to further explore the efficacy and safety of Fruquintinib combined with S-1 in treating recurrent or metastatic esophageal squamous cell carcinoma after the failure of conventional treatments.

DETAILED DESCRIPTION:
Esophageal cancer is one of the most common malignant tumor and esophageal squamous cell carcinoma is the main pathological type of esophageal carcinoma in China. Among patients with advanced or metastatic esophageal squamous cell carcinoma, the addition of immunotherapy to chemotherapy, compared with placebo and chemotherapy, significantly improved overall survival and progression-free survival.Treatment of recurrent or metastatic esophageal squamous cell carcinoma is usually poor. New treatments were needed. Fruquintinib is an orally antiangiogenic agents, which target VEGFR1/2/3. A combination of Fruquintinib and s-1 for advanced or metastatic esophageal squamous cell carcinoma could be a novel therapy. Therefore, investigators initialize this phase II study to explore the safety of fruquintinib and S-1 combination treatment in ESCC patients with after failure in 1st-line immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, age:≥18 years old
* Imageology diagnosed with refractory or metastatic esophageal squamous cell carcinoma
* Disease progression after the last dose of the first-line therapy (with immunotherapy, without fluoropyrimidine)
* At least one measurable lesion (RECIST1.1)
* Good performance status Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0 to 2
* Life expectancy of more than 12 weeks
* The test value for bone marrow, liver and renal function evaluation within 7 days prior to first dosing should meet requirements
* Negative of blood pregnancy test within 7 days prior to first dosing for fertile female patients. Fertile female and male patients agree to use effective contraceptive methods during the study and within 6 months post to the last dose, such as double barrier contraception, condoms, oral or injection contraceptives, intrauterine devices, abstinence, etc. All female patients will be considered fertile unless the female patient has natural menopause or has undergone artificial menopause or sterilization (hysterectomy, bilateral appendage resection);
* Signed informed consent

Exclusion Criteria:

* Absolute neutrophil count (ANC) <1.5×109/L, platelet count <75×109/L, and hemoglobin <9g/dL
* Serum total bilirubin >1.5× the upper limit of normal (ULN)
* Alanine aminotransferase (ALT)/aspartate aminotransferase (AST) >2.5×ULN
* Creatinine > 1.5 × ULN or creatinine clearance <50 mL/min
* Activated partial thromboplastin time (APTT)> 1.5 × ULN
* The investigators determined clinically significant severe electrolyte abnormalities.
* Proteinuria ≥ 2+ (1.0g/24hr)
* Drug uncontrollable hypertension, defined as systolic blood pressure ≥ 140 mmHg and / or diastolic blood pressure ≥ 90 mmHg
* The patients have active ulcer of stomach and duodenum, ulcerative colitis and other digestive tract diseases or unresectable tumors with active bleeding, or other conditions that may cause gastrointestinal bleeding and perforation, as judged by investigators; or the existence of gastrointestinal perforation or gastrointestinal fistula uncured post to previous surgical treatment
* Patients with evidence or history of propensity to hemorrhage within 2 months prior to first dosing, regardless of severity(such as melena, hematemesis, hemoptysis, bloody stools）
* Arterial thrombosis or deep venous thrombosis within 6 months prior to first dosing, or thromboembolic events
* Cardiovascular diseases of significant clinical significance, including, but not limited to acute myocardial infarction, severe/unstable angina pectoris or coronary artery bypass grafting within 6 months prior to first dosing, congestive heart failure with New York Heart Association (NYHA) grade ≥ 2; Left ventricular ejection fraction (LVEF) < 50%
* Uncontrolled malignant pleural effusion, ascites or pericardial effusion
* Previous treatment with anti-vascular endothelial growth factor receptor (VEGFR) inhibitors
* A history of other malignancies within 5 years prior to inclusion, except for cervical carcinoma in situ, basal or squamous cell skin cancer
* Distal metastasis to brain
* History of clinically significant hepatic disease, including, but not limited to, known hepatitis B virus (HBV) infection with HBV DNA positive (copies ≥1×104/ml); known hepatitis C virus infection with HCV RNA positive
* Women who are pregnant or lactating
* Patients considered unsuitable for inclusion in this study by the investigator
* Patients considered a serious mental or mental abnormality

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2022-03-30 (Actual); Primary Completion 2024-03-30 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | From date of first dose of study drug until disease progression, withdrawal of consent, death (up to approximately 1 year)
  PFS defined as the time from the date of randomization to the first evidence of disease progression as defined by response evaluation criteria in solid tumors (RECIST) v1.1 or death from any cause.

SECONDARY OUTCOMES:
Overall survival (OS) | Baseline to measured date of death from any cause (up to approximately 1 year)
Objective response rate (ORR) | from treatment up to progressive disease or EOT due to any cause up to 1 year
  Tumor assessment will be performed using radiography method every 6 weeks until the occurrence of progressive disease (PD), using RECIST v 1.1
Disease control rate (DCR) | from treatment up to progressive disease or EOT due to any cause up to 1 year
  Tumor assessment will be performed using radiography method every 6 weeks until the occurrence of progressive disease (PD), using RECIST v 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Zhao Lin, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No